CLINICAL TRIAL: NCT01447446
Title: Non-Interventional Cohort Study on the Utilization and Impact of Dual and Triple Therapies Based on Pegylated Interferon for the Treatment of Chronic Hepatitis C
Brief Title: An Observational Study on Dual And Triple Therapies Based on Peginterferon Alfa (e.g. Pegasys) in Patients With Chronic Hepatitis C
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: MV25599
Record Dates: First submitted 2011-10-04; First posted 2011-10-06 (Estimated); Results first posted 2017-03-30 (Actual); Last update posted 2017-03-30 (Actual); Status verified 2016-12

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2a; peginterferon alfa-2b; Ribavirin; N-(3-amino-1-(cyclobutylmethyl)-2,3-dioxopropyl)-3-(2-((((1,1-dimethylethyl)amino)carbonyl)amino)-3,3-dimethyl-1-oxobutyl)-6,6-dimethyl-3-azabicyclo(3.1.0)hexan-2-carboxamide; telaprevir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (6):
- Dual Therapy: Peg-IFN Alfa-2a + Ribavirin: Participants with chronic hepatitis C (CHC) receiving dual therapy (pegylated interferon alfa-2a [peg-IFN Alfa-2a] along with ribavirin according to standard of care and in line with local labeling) were followed up for the duration of their treatment and for up to 24 weeks after therapy.
  Interventions: Drug: Peg-IFN Alfa-2a; Drug: Ribavirin
- Dual Therapy: Peg-IFN Alfa-2b + Ribavirin: Participants with CHC receiving dual therapy (pegylated interferon alfa-2b [peg-IFN Alfa-2b] along with ribavirin according to standard of care and in line with local labeling) were followed for the duration of their treatment and for up to 24 weeks after therapy.
  Interventions: Drug: Peg-IFN Alfa-2b; Drug: Ribavirin
- Triple Therapy: Boceprevir + Peg-IFN Alfa-2a + Ribavirin: Participants with CHC receiving triple therapy (peg-IFN Alfa-2a along with ribavirin and boceprevir according to standard of care and in line with local labeling) were followed for the duration of their treatment and for up to 24 weeks after therapy.
  Interventions: Drug: Peg-IFN Alfa-2a; Drug: Ribavirin; Drug: Boceprevir
- Triple Therapy: Boceprevir + Peg-IFN Alfa-2b + Ribavirin: Participants with CHC receiving triple therapy (peg-IFN Alfa-2b along with ribavirin and boceprevir according to standard of care and in line with local labeling) were followed for the duration of their treatment and for up to 24 weeks after therapy.
  Interventions: Drug: Peg-IFN Alfa-2b; Drug: Ribavirin; Drug: Boceprevir
- Triple Therapy: Telaprevir + Peg-IFN Alfa-2a + Ribavirin: Participants with CHC receiving triple therapy (peg-IFN Alfa-2a along with ribavirin and telaprevir according to standard of care and in line with local labeling) were followed for the duration of their treatment and for up to 24 weeks after therapy.
  Interventions: Drug: Peg-IFN Alfa-2a; Drug: Ribavirin; Drug: Telaprevir
- Triple Therapy: Telaprevir + Peg-IFN Alfa-2b + Ribavirin: Participants with CHC receiving triple therapy (peg-IFN Alfa-2b along with ribavirin and telaprevir according to standard of care and in line with local labeling) were followed for the duration of their treatment and for up to 24 weeks after therapy.
  Interventions: Drug: Peg-IFN Alfa-2b; Drug: Ribavirin; Drug: Telaprevir

INTERVENTIONS:
Drug: Peg-IFN Alfa-2a — Peg-IFN Alfa-2a according to standard of care and in line with local labeling.
  Groups: Dual Therapy: Peg-IFN Alfa-2a + Ribavirin; Triple Therapy: Boceprevir + Peg-IFN Alfa-2a + Ribavirin; Triple Therapy: Telaprevir + Peg-IFN Alfa-2a + Ribavirin
Drug: Peg-IFN Alfa-2b — Peg-IFN Alfa-2b according to standard of care and in line with local labeling.
  Groups: Dual Therapy: Peg-IFN Alfa-2b + Ribavirin; Triple Therapy: Boceprevir + Peg-IFN Alfa-2b + Ribavirin; Triple Therapy: Telaprevir + Peg-IFN Alfa-2b + Ribavirin
Drug: Ribavirin — Ribavirin according to standard of care and in line with local labeling.
Drug: Boceprevir — Boceprevir according to standard of care and in line with local labeling.
  Groups: Triple Therapy: Boceprevir + Peg-IFN Alfa-2a + Ribavirin; Triple Therapy: Boceprevir + Peg-IFN Alfa-2b + Ribavirin
Drug: Telaprevir — Telaprevir according to standard of care and in line with local labeling.
  Groups: Triple Therapy: Telaprevir + Peg-IFN Alfa-2a + Ribavirin; Triple Therapy: Telaprevir + Peg-IFN Alfa-2b + Ribavirin

SUMMARY:
This prospective, multicenter, observational cohort study will evaluate the efficacy and safety of pegylated interferon alfa (peginterferon alfa) (e.g. Pegasys) plus ribavirin and treatment regimens containing direct-acting antivirals in participants with chronic hepatitis C who are treatment-naïve or treatment-experienced and HIV HCV co-infected. Data will be collected from participants receiving treatment according to current Summary of Product Characteristics (SPC) and local labeling for the duration of their treatment and a 24-week follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Adult (according to local legislation) participants
* Chronic hepatitis C (HCV)
* Naive or treatment experienced, HIV-HCV co-infected or HCV mono-infected
* Receiving treatment for HCV with pegylated interferons plus ribavirin or regimens containing direct-acting antivirals (DAA) according to standard of care and in line with current SPC/local labeling

Exclusion Criteria:

* Contraindications according to SPC/local labeling
* Treatment started >4 weeks before entering study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic hepatitis C (CHC) participants (naïve or treatment experienced, including HIV HCV co-infected) receiving combination therapy with pegylated interferons plus ribavirin or treatment regimens containing direct-acting antivirals.
Sampling Method: Probability Sample
Enrollment: 4442 (Actual)
Dates: Start 2011-09; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (215):
- Belgium (17):
  - Antwerp
  - Bouge
  - Brussels
  - Edegem
  - Ghent
  - Gilly (Charleroi)
  - Hasselt
  - Heusy
  - Kortrijk
  - Leuven
  - Liège
  - Mons
  - Montignies-sur-Sambre
  - Namur
  - Ostend
  - Roeselare
  - Verviers
- Egypt (4):
  - Alexandria
  - Cairo
  - Giza
  - Tanta
- Estonia (4):
  - Kohtla-Järve
  - Pärnu
  - Tallinn
  - Tartu
- France (53):
  - Aix-en-Provence
  - Amiens
  - Argenteuil
  - Avignon
  - Besançon
  - Béziers
  - Boulogne-Billancourt
  - Bourgoin
  - Caen
  - Chambray-lès-Tours
  - Clichy
  - Creil
  - Créteil
  - Épinay-sur-Seine
  - Évry
  - Freyming-Merlebach
  - Gonesse
  - Grasse
  - Hyères
  - La Tronche
  - Lagny-sur-Marne
  - Lille
  - Limoges
  - Lomme
  - Lyon
  - Mantes-la-Jolie
  - Marseille
  - Meaux
  - Montpellier
  - Nice
  - Nîmes
  - Orange
  - Orléans
  - Paris
  - Pau
  - Perpignan
  - Pessac
  - Reims
  - Rennes
  - Rouen
  - Saint-Laurent-du-Var
  - Saint-Nazaire
  - Saint-Priest-en-Jarez
  - Strasbourg
  - Suresnes
  - Toulon
  - Toulouse
  - Tourcoing
  - Vandœuvre-lès-Nancy
  - Vannes
  - Villejuif
  - Villeneuve Maguelone
  - Villeneuve-Saint-Georges
- Germany (14):
  - Aachen
  - Berlin
  - Burghausen
  - Cologne
  - Düsseldorf
  - Erlangen
  - Essen
  - Kassel
  - Lübeck
  - Magdeburg
  - Mannheim
  - Rostock
  - Rottenburg
  - Tübingen
- Greece (7):
  - Alexandroupoli
  - Athens
  - Ioannina
  - Larissa
  - Nea Kifissia
  - Pátrai
  - Thessaloniki
- Hungary (18):
  - Ajka
  - Balassagyarmat
  - Békéscsaba
  - Budapest
  - Debrecen
  - Gyula
  - Kaposvár
  - Kecskemét
  - Miskolc
  - Nyíregyháza
  - Pécs
  - Sopron
  - Szeged
  - Székesfehérvár
  - Szolnok
  - Szombathely
  - Tatabánya
  - Zalaegerszeg
- Dublin, Ireland
- Italy (35):
  - Chieti, Abruzzo
  - Bari, Apulia
  - Bisceglie, Apulia
  - Castellana Grotte, Apulia
  - San Giovanni Rotondo, Apulia
  - Reggio Calabria, Calabria
  - Avellino, Campania
  - Gragnano, Campania
  - Marcianise, Campania
  - Napoli, Campania
  - Nocera Inferiore, Campania
  - Nola, Campania
  - Bologna, Emilia-Romagna
  - Modena, Emilia-Romagna
  - Parma, Emilia-Romagna
  - Piacenza, Emilia-Romagna
  - Udine, Friuli Venezia Giulia
  - Rome, Lazio
  - Genoa, Liguria
  - Savona, Liguria
  - Busto Arsizio, Lombardy
  - Milan, Lombardy
  - Biella, Piedmont
  - Cuorgnè (TO), Piedmont
  - Omegna (VB), Piedmont
  - Cagliari, Sardinia
  - Sassari, Sardinia
  - Catania, Sicily
  - Messina, Sicily
  - Palermo, Sicily
  - Torrette Di Ancona, The Marches
  - Arezzo, Tuscany
  - Florence, Tuscany
  - Livorno, Tuscany
  - Padua, Veneto
- Safat, Kuwait
- Lebanon (4):
  - Baabda
  - Beirut
  - Nabatieh
  - Tripoli
- Morocco (4):
  - Casablanca
  - Fes
  - Marrakesh
  - Rabat
- Skopje, North Macedonia
- Muscat, Oman
- Pakistan (5):
  - Faisalabad
  - Gujranwala
  - Karachi
  - Lahore
  - Rawalpindi
- Portugal (8):
  - Almada
  - Amadora
  - Aveiro
  - Beja
  - Coimbra
  - Faro
  - Lisbon
  - Porto
- Doha, Qatar
- Romania (5):
  - Bucharest
  - Cluj-Napoca
  - Constanța
  - Iași
  - Timișoara
- Saudi Arabia (2):
  - Holy Makkah
  - Riyadh
- Serbia (2):
  - Belgrade
  - Novi Sad
- Sweden (3):
  - Gävle
  - Karlstad
  - Uppsala
- Switzerland (2):
  - Lugano
  - Sankt Gallen
- Aleppo, Syria
- Taiwan (4):
  - Kaohsiung City
  - Taichung
  - Taipei
  - Taoyuan District
- Turkey (Türkiye) (10):
  - Adana
  - Ankara
  - Hatay
  - Istanbul
  - ISTANBULt
  - Izmir
  - Kayseri
  - Mersin
  - Tokat Province
  - Trabzon
- United Arab Emirates (3):
  - Al Ain City
  - Dubai
  - Sharjah city
- United Kingdom (5):
  - Dundee
  - Hull
  - London
  - Manchester
  - Nottingham

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 4442 participants were enrolled in the study, one participant had double enrollment. Out of 4442 participants, analyses were restricted to only core population, which included 4100 participants.
Groups:
- Dual Therapy: Peg-IFN Alfa-2a + Ribavirin: Participants with CHC receiving dual therapy (pegylated interferon alfa-2a [peg-IFN Alfa-2a] along with ribavirin according to standard of care and in line with local labeling) were followed for the duration of their treatment and for up to 24 weeks after therapy.
Period: Overall Study
Arm/Group | Dual Therapy: Peg-IFN Alfa-2a + Ribavirin | Dual Therapy: Peg-IFN Alfa-2b + Ribavirin | Triple Therapy: Boceprevir + Peg-IFN Alfa-2a + Ribavirin | Triple Therapy: Boceprevir + Peg-IFN Alfa-2b + Ribavirin | Triple Therapy: Telaprevir + Peg-IFN Alfa-2a + Ribavirin | Triple Therapy: Telaprevir + Peg-IFN Alfa-2b + Ribavirin
Started | 2312 (Started means participants who started treatment and included in core population.) | 496 | 292 | 93 | 821 | 86
Completed | 1590 (Completed means the participants who completed the 24- weeks of follow-up period.) | 331 (Insuff.=Insufficient VR= Virological response TRT.=Treatment SVR= Sustained Virological Response) | 192 | 60 | 610 | 54
Not Completed | 722 | 165 | 100 | 33 | 211 | 32
Not completed — Death | 6 | 3 | 2 | 1 | 7 | 0
Not completed — Adverse Event | 3 | 0 | 1 | 0 | 2 | 0
Not completed — Failure to Return/Consent Withdrawn | 357 | 78 | 31 | 7 | 69 | 9
Not completed — Insuff. VR/TRT too Short to Expect VR | 300 | 71 | 52 | 21 | 92 | 14
Not completed — Administrative/Other | 34 | 9 | 10 | 2 | 33 | 4
Not completed — SVR12 Assessment | 13 | 1 | 2 | 1 | 5 | 5
Not completed — New Treatment Started | 8 | 2 | 1 | 0 | 2 | 0
Not completed — Reason not Specified | 1 | 1 | 1 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Core population: treatment-naive/experienced participants who were without contraindication to Peg-IFN and RBV, end stage renal disease, major organ transplantation, co-infection with hepatitis B or HIV, acute hepatitis and with positive HCV RNA at baseline, known genotype, 1 of 6 treatment (excluding non-G1 participants receiving triple therapy).
Groups:
- Dual Therapy: Peg-IFN Alfa-2a + Ribavirin: Participants with CHC receiving dual therapy (peg-IFN Alfa-2a along with ribavirin according to standard of care and in line with local labeling) were followed for the duration of their treatment and for up to 24 weeks after therapy.
- Dual Therapy: Peg-IFN Alfa-2b + Ribavirin: Participants with CHC receiving dual therapy (peg-IFN Alfa-2b along with ribavirin according to standard of care and in line with local labeling) were followed for the duration of their treatment and for up to 24 weeks after therapy.
- Total: Total of all reporting groups
Arm/Group | Dual Therapy: Peg-IFN Alfa-2a + Ribavirin | Dual Therapy: Peg-IFN Alfa-2b + Ribavirin | Triple Therapy: Boceprevir + Peg-IFN Alfa-2a + Ribavirin | Triple Therapy: Boceprevir + Peg-IFN Alfa-2b + Ribavirin | Triple Therapy: Telaprevir + Peg-IFN Alfa-2a + Ribavirin | Triple Therapy: Telaprevir + Peg-IFN Alfa-2b + Ribavirin | Total
Number analyzed (Participants) | 2312 | 496 | 292 | 93 | 821 | 86 | 4100
Age, Customized [Number; unit: participants]
  Less Than or Equal to (<=) 45 Years | 987 | 178 | 73 | 21 | 184 | 14 | 1457
  Greater (>) 45 years | 1325 | 318 | 219 | 72 | 637 | 72 | 2643
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 910 | 250 | 108 | 37 | 331 | 43 | 1679
  Male | 1402 | 246 | 184 | 56 | 490 | 43 | 2421

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virological Response at 24 Weeks Post Completion of the Treatment Period (SVR24)
Description: SVR24 rate for dual therapy participants is defined as percentage of participants with hepatitis C virus (HCV) ribonucleic acid (RNA) less than (<) 50 international unit/milliliters (IU/mL) (as measured by a commercially available HCV RNA test with lower limit of detection less than or equal to [<=] 50 IU/mL) at 24 weeks post completion of the treatment period. If a quantitative test was used, the lower limit of quantification had to be <=50 IU/mL. SVR24 for triple therapy participants is defined as percentage of participants with undetectable HCV RNA assessed by a test with lower limit of detection <= 50 IU/mL at 24 weeks post completion of the treatment period.
Time Frame: 24 weeks after end of treatment (up to 118 weeks)
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dual Therapy: Peg-IFN Alfa-2a + Ribavirin | Dual Therapy: Peg-IFN Alfa-2b + Ribavirin | Triple Therapy: Boceprevir + Peg-IFN Alfa-2a + Ribavirin | Triple Therapy: Boceprevir + Peg-IFN Alfa-2b + Ribavirin | Triple Therapy: Telaprevir + Peg-IFN Alfa-2a + Ribavirin | Triple Therapy: Telaprevir + Peg-IFN Alfa-2b + Ribavirin
Number analyzed (Participants) | 2312 | 496 | 292 | 93 | 821 | 86
percentage of participants | 52.1 [50.1 to 54.2] | 49.4 [44.9 to 53.9] | 46.6 [40.7 to 52.5] | 50.5 [40.0 to 61.1] | 57.7 [54.3 to 61.1] | 47.7 [36.8 to 58.7]

2. Primary Outcome: Percentage of Participants With Sustained Virological Response at 12 Weeks Post Completion of the Treatment Period (SVR12)
Description: SVR12 rate for dual therapy participants is defined as percentage of participants with hepatitis C virus (HCV) ribonucleic acid (RNA) less than (<) 50 international unit/milliliters (IU/mL) (as measured by a commercially available HCV RNA test with lower limit of detection less than or equal to [<=] 50 IU/mL) at 12 weeks post completion of the treatment period. If a quantitative test was used, the lower limit of quantification had to be <=50 IU/mL. SVR12 for triple therapy participants is defined as percentage of participants with undetectable HCV RNA assessed by a test with lower limit of detection <= 50 IU/mL at 12 weeks post completion of the treatment period.
Time Frame: 12 weeks after end of treatment (up to 118 weeks)
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dual Therapy: Peg-IFN Alfa-2a + Ribavirin | Dual Therapy: Peg-IFN Alfa-2b + Ribavirin | Triple Therapy: Boceprevir + Peg-IFN Alfa-2a + Ribavirin | Triple Therapy: Boceprevir + Peg-IFN Alfa-2b + Ribavirin | Triple Therapy: Telaprevir + Peg-IFN Alfa-2a + Ribavirin | Triple Therapy: Telaprevir + Peg-IFN Alfa-2b + Ribavirin
Number analyzed (Participants) | 2312 | 496 | 292 | 93 | 821 | 86
percentage of participants | 54.3 [52.2 to 56.3] | 51.0 [46.5 to 55.5] | 50.0 [44.1 to 55.9] | 53.8 [43.1 to 64.2] | 62.0 [58.6 to 65.3] | 57.0 [45.8 to 67.6]

3. Secondary Outcome: Virological Response at Various on Treatment Time Points and End of Treatment (EOT)
Description: Virological response (VR) for dual therapy participants is defined as HCV RNA <50 IU/mL as assessed by a qualitative HCV RNA test with a lower limit of detection (LLD) <=50 IU/mL or as assessed by a quantitative test with a lower limit of quantification (LLQ) <=50 IU/mL for all time points concerned. Results of HCV RNA tests with LLD and LLQ >50 IU/mL were considered as non-response. VR for triple therapy participants is defined as undetectable HCV RNA assessed by a test with lower limit of detection <=50 IU/mL (UVR). Results of HCV RNA tests with an LLD >50 IU/mL were considered as non-response for triple therapy participants.
Time Frame: Week 4, 12 and End of treatment (EOT) (up to 96 weeks)
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dual Therapy: Peg-IFN Alfa-2a + Ribavirin | Dual Therapy: Peg-IFN Alfa-2b + Ribavirin | Triple Therapy: Boceprevir + Peg-IFN Alfa-2a + Ribavirin | Triple Therapy: Boceprevir + Peg-IFN Alfa-2b + Ribavirin | Triple Therapy: Telaprevir + Peg-IFN Alfa-2a + Ribavirin | Triple Therapy: Telaprevir + Peg-IFN Alfa-2b + Ribavirin
Number analyzed (Participants) | 2312 | 496 | 292 | 93 | 821 | 86
percentage of participants
  VR by Week 4 | 39.5 [37.5 to 41.5] | 40.1 [35.8 to 44.6] | 9.9 [6.8 to 14.0] | 9.7 [4.5 to 17.6] | 49.8 [46.3 to 53.3] | 51.2 [40.1 to 62.1]
  VR by Week 12 | 71.3 [69.4 to 73.2] | 67.7 [63.4 to 71.8] | 56.8 [51.0 to 62.6] | 59.1 [48.5 to 69.2] | 80.8 [77.9 to 83.4] | 73.3 [62.6 to 82.2]
  VR by EOT | 73.6 [71.7 to 75.4] | 70.6 [66.3 to 74.5] | 67.1 [61.4 to 72.5] | 72.0 [61.8 to 80.9] | 74.9 [71.8 to 77.8] | 66.3 [55.3 to 76.1]

4. Secondary Outcome: Virological Relapse After End of Treatment
Description: Virological relapse defined as non-virological response (non-VR)/non-undetectable virological response (non-UVR) at the last HCV RNA assessment during the treatment-free follow-up period in participants with VR/UVR at EOT. Here, number of participants analyzed is the participants with end of treatment response (EoT-R) who also had an HCV RNA test at least 12 weeks after EoT or whose last follow-up HCV RNA test showed non-response (HCV RNA >=50 IU/mL).
Time Frame: Up to 24 weeks after EOT (up to 118 weeks)
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dual Therapy: Peg-IFN Alfa-2a + Ribavirin | Dual Therapy: Peg-IFN Alfa-2b + Ribavirin | Triple Therapy: Boceprevir + Peg-IFN Alfa-2a + Ribavirin | Triple Therapy: Boceprevir + Peg-IFN Alfa-2b + Ribavirin | Triple Therapy: Telaprevir + Peg-IFN Alfa-2a + Ribavirin | Triple Therapy: Telaprevir + Peg-IFN Alfa-2b + Ribavirin
Number analyzed (Participants) | 1521 | 314 | 181 | 63 | 581 | 53
percentage of participants | 18.4 [16.5 to 20.4] | 19.7 [15.5 to 24.6] | 21.0 [15.3 to 27.7] | 20.6 [11.5 to 32.7] | 13.8 [11.1 to 16.8] | 7.5 [2.1 to 18.2]

5. Secondary Outcome: Virological Breakthrough
Description: Virological breakthrough/rebound defined as non-VR/non-UVR during the treatment period (including end of treatment) in participants with prior VR/UVR or an increase of HCV RNA by >=1 log10 during the treatment period in comparison to the lowest HCV RNA (nadir) previously measured during the treatment period in participants without VR/UVR during the treatment period. Here, Number of participants analyzed is the participants with at least 2 on-treatment HCV RNA assessments (including EoT) or 1 on-treatment HCV RNA assessment (excluding EoT) and response at EoT by backward imputation.
Time Frame: Up to EOT (up to 118 weeks)
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dual Therapy: Peg-IFN Alfa-2a + Ribavirin | Dual Therapy: Peg-IFN Alfa-2b + Ribavirin | Triple Therapy: Boceprevir + Peg-IFN Alfa-2a + Ribavirin | Triple Therapy: Boceprevir + Peg-IFN Alfa-2b + Ribavirin | Triple Therapy: Telaprevir + Peg-IFN Alfa-2a + Ribavirin | Triple Therapy: Telaprevir + Peg-IFN Alfa-2b + Ribavirin
Number analyzed (Participants) | 2079 | 437 | 275 | 88 | 785 | 74
percentage of participants | 5.4 [4.5 to 6.4] | 4.8 [3.0 to 7.3] | 8.7 [5.7 to 12.7] | 15.9 [9.0 to 25.2] | 15.0 [12.6 to 17.7] | 21.6 [12.9 to 32.7]

6. Secondary Outcome: Percentage of Participants With Sustained Virological Response (SVR) in Participants With Dose Reductions or Treatment Interruptions
Description: SVR 12 and 24 rates for dual therapy participants are defined as percentage of participants with hepatitis C virus (HCV) ribonucleic acid (RNA) less than (<) 50 international unit/milliliters (IU/mL) (as measured by a commercially available HCV RNA test with lower limit of detection less than or equal to [<=] 50 IU/mL) at 12 or 24 weeks post completion of the treatment period. If a qualitative test was used, then the lower limit of detection has to be <=50 IU/mL. SVR12 and 24 rates for triple therapy participants are defined as percentage of participants with undetectable HCV RNA assessed by a test with lower limit of detection <= 50 IU/mL at 12 or 24 weeks post completion of the treatment period. Here, number of participants analyzed excluded the participants with premature withdrawal due to lack of efficacy or non-safety reasons and participants without dose reductions or interruptions during the first 99 study days.
Time Frame: Up to first 12 weeks of treatment
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dual Therapy: Peg-IFN Alfa-2a + Ribavirin | Dual Therapy: Peg-IFN Alfa-2b + Ribavirin | Triple Therapy: Boceprevir + Peg-IFN Alfa-2a + Ribavirin | Triple Therapy: Boceprevir + Peg-IFN Alfa-2b + Ribavirin | Triple Therapy: Telaprevir + Peg-IFN Alfa-2a + Ribavirin | Triple Therapy: Telaprevir + Peg-IFN Alfa-2b + Ribavirin
Number analyzed (Participants) | 116 | 33 | 29 | 7 | 79 | 9
percentage of participants
  SVR at Week 12 After EOT | 37.1 [28.3 to 46.5] | 27.3 [13.3 to 45.5] | 20.7 [8.0 to 39.7] | 14.3 [0.4 to 57.9] | 35.4 [25.0 to 47.0] | 44.4 [13.7 to 78.8]
  SVR at Week 24 EOT | 35.3 [26.7 to 44.8] | 24.2 [11.1 to 42.3] | 17.2 [5.8 to 35.8] | 14.3 [0.4 to 57.9] | 34.2 [23.9 to 45.7] | 44.4 [13.7 to 78.8]

7. Secondary Outcome: Percentage of Participants With Very Rapid Virological Response, Rapid Virological Response, Complete Early Virological Response and Partial Early Virological Response (pEVR) During First 12 Weeks
Description: Percentage of participants with very rapid virological response (VRVR) (defined as VR/UVR by study week 2), rapid virological response (RVR) (defined as VR/UVR by study week 4, but no VRVR), complete early virological response (cEVR) (defined as VR/UVR by study week 12, but no VRVR or RVR) and partial early virological response (pEVR) (defined as a 2 log10 drop of HCV RNA by study week 12, but no VRVR, RVR or cEVR) were reported.
Time Frame: Up to 12 weeks
Population: The data for all of the above mentioned virological responses were not collected and was not analyzed.
Arm/Group | Dual Therapy: Peg-IFN Alfa-2a + Ribavirin | Dual Therapy: Peg-IFN Alfa-2b + Ribavirin | Triple Therapy: Boceprevir + Peg-IFN Alfa-2a + Ribavirin | Triple Therapy: Boceprevir + Peg-IFN Alfa-2b + Ribavirin | Triple Therapy: Telaprevir + Peg-IFN Alfa-2a + Ribavirin | Triple Therapy: Telaprevir + Peg-IFN Alfa-2b + Ribavirin
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Percentage of Participants Achieving Extended (Rapid) Virological Response (eRVR)
Description: Extended (rapid) virological response (eRVR) defined as UVR at weeks 4 and 12 for telaprevir, and as UVR at weeks 8 and 24 for boceprevir.
Time Frame: Up to 98 weeks
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Triple Therapy: Boceprevir + Peg-IFN Alfa-2a + Ribavirin | Triple Therapy: Boceprevir + Peg-IFN Alfa-2b + Ribavirin | Triple Therapy: Telaprevir + Peg-IFN Alfa-2a + Ribavirin | Triple Therapy: Telaprevir + Peg-IFN Alfa-2b + Ribavirin
Number analyzed (Participants) | 292 | 93 | 821 | 86
percentage of participants | 37.7 [32.1 to 43.5] | 32.3 [22.9 to 42.7] | 45.6 [42.1 to 49.0] | 47.7 [36.8 to 58.7]

9. Secondary Outcome: Duration of Overall Treatment
Description: Duration of overall treatment was defined as the time between first and last administration of any study drug, in weeks.
Time Frame: Up to 118 weeks
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | Dual Therapy: Peg-IFN Alfa-2a + Ribavirin | Dual Therapy: Peg-IFN Alfa-2b + Ribavirin | Triple Therapy: Boceprevir + Peg-IFN Alfa-2a + Ribavirin | Triple Therapy: Boceprevir + Peg-IFN Alfa-2b + Ribavirin | Triple Therapy: Telaprevir + Peg-IFN Alfa-2a + Ribavirin | Triple Therapy: Telaprevir + Peg-IFN Alfa-2b + Ribavirin
Number analyzed (Participants) | 2312 | 496 | 292 | 93 | 821 | 86
Weeks | 34.2 (16.04) | 31.3 (15.73) | 35.2 (17.48) | 35.3 (15.27) | 33.2 (15.03) | 31.2 (15.95)

10. Secondary Outcome: Percentage of Participants Treated According to Label/Summary of Product Characteristics (SPC)
Time Frame: Up to 118 weeks
Population: The data for this outcome measure were not collected and analyzed because the standard of care has changed significantly since the development of the study protocol, this comparison was no longer of practical value.
Arm/Group | Dual Therapy: Peg-IFN Alfa-2a + Ribavirin | Dual Therapy: Peg-IFN Alfa-2b + Ribavirin | Triple Therapy: Boceprevir + Peg-IFN Alfa-2a + Ribavirin | Triple Therapy: Boceprevir + Peg-IFN Alfa-2b + Ribavirin | Triple Therapy: Telaprevir + Peg-IFN Alfa-2a + Ribavirin | Triple Therapy: Telaprevir + Peg-IFN Alfa-2b + Ribavirin
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

11. Secondary Outcome: Percentage of Participants Who Discontinued Treatment With PEG-IFN and Ribavirin (RBV)
Description: Participants who prolonged the treatment period from 72 weeks were not reported.
Time Frame: Up to 72 weeks of treatment
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Dual Therapy: Peg-IFN Alfa-2a + Ribavirin | Dual Therapy: Peg-IFN Alfa-2b + Ribavirin | Triple Therapy: Boceprevir + Peg-IFN Alfa-2a + Ribavirin | Triple Therapy: Boceprevir + Peg-IFN Alfa-2b + Ribavirin | Triple Therapy: Telaprevir + Peg-IFN Alfa-2a + Ribavirin | Triple Therapy: Telaprevir + Peg-IFN Alfa-2b + Ribavirin
Number analyzed (Participants) | 2312 | 496 | 292 | 93 | 821 | 86
percentage of participants
  Discontinued PEG-IFN During Week 1 to Week 12 | 5.7 | 8.3 | 9.2 | 9.7 | 9.9 | 11.6
  Discontinued RBV During Week 1 to Week 12 | 6.3 | 9.1 | 9.6 | 10.8 | 10.8 | 12.8
  Discontinued PEG-IFN During Week 13 to Week 24 | 13.5 | 17.1 | 16.8 | 14.0 | 10.2 | 12.8
  Discontinued RBV During Week 13 to Week 24 | 22.1 | 22.4 | 17.1 | 16.1 | 13.9 | 19.8
  Discontinued PEG-IFN During Week 25 to Week 48 | 41.7 | 41.3 | 30.1 | 29.0 | 41.0 | 43.0
  Discontinued RBV During Week 25 to Week 48 | 43.0 | 46.6 | 41.1 | 41.9 | 44.9 | 41.9
  Discontinued PEG-IFN During Week 49 to Week 72 | 36.2 | 32.1 | 41.1 | 47.3 | 38.9 | 32.6
  Discontinued RBV During Week 49 to Week 72 | 26.6 | 21.0 | 29.1 | 31.2 | 30.3 | 25.6

12. Secondary Outcome: Percentage of Participants Who Discontinued Treatment With Direct-Acting Anti-viral (DAA)
Description: Participants who prolonged the treatment period from 72 weeks were not reported. Participants who discontinued their treatment as planned were included. Here, number of participant analyzed is the total number of participants who received direct-acting anti-viral (DAA).
Time Frame: Up to 72 weeks of treatment
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Triple Therapy: Boceprevir + Peg-IFN Alfa-2a + Ribavirin | Triple Therapy: Boceprevir + Peg-IFN Alfa-2b + Ribavirin | Triple Therapy: Telaprevir + Peg-IFN Alfa-2a + Ribavirin | Triple Therapy: Telaprevir + Peg-IFN Alfa-2b + Ribavirin
Number analyzed (Participants) | 292 | 93 | 821 | 86
percentage of participants
  Discontinued DAA During Week 1 to Week 2 | 6.8 | 7.5 | 1.7 | 4.7
  Discontinued DAA During Week 3 to Week 4 | 2.1 | 1.1 | 1.5 | 4.7
  Discontinued DAA During Week 5 to Week 12 | 13.4 | 8.6 | 24.7 | 22.1
  Discontinued DAA During Week 13 to Week 24 | 16.1 | 18.3 | 71.7 | 68.6
  Discontinued DAA During Week 25 to Week 48 | 59.2 | 64.5 | 0.4 | 0.0

13. Secondary Outcome: Percentage of Participants With Concomitant Medical Condition at Baseline
Time Frame: Baseline
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Dual Therapy: Peg-IFN Alfa-2a + Ribavirin | Dual Therapy: Peg-IFN Alfa-2b + Ribavirin | Triple Therapy: Boceprevir + Peg-IFN Alfa-2a + Ribavirin | Triple Therapy: Boceprevir + Peg-IFN Alfa-2b + Ribavirin | Triple Therapy: Telaprevir + Peg-IFN Alfa-2a + Ribavirin | Triple Therapy: Telaprevir + Peg-IFN Alfa-2b + Ribavirin
Number analyzed (Participants) | 2312 | 496 | 292 | 93 | 821 | 86
percentage of participants | 48.1 | 50.4 | 65.8 | 68.8 | 67.2 | 41.9

14. Secondary Outcome: Percentage of Participants With Adverse Events (AE)
Description: An AE was defined as any adverse medical event that occurred after the participant used the investigational medicinal product (IMP) or other intervention behaviors specified by the protocol in the clinical trial regardless of relationship to the study treatment.
Time Frame: Up to 118 weeks
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Dual Therapy: Peg-IFN Alfa-2a + Ribavirin | Dual Therapy: Peg-IFN Alfa-2b + Ribavirin | Triple Therapy: Boceprevir + Peg-IFN Alfa-2a + Ribavirin | Triple Therapy: Boceprevir + Peg-IFN Alfa-2b + Ribavirin | Triple Therapy: Telaprevir + Peg-IFN Alfa-2a + Ribavirin | Triple Therapy: Telaprevir + Peg-IFN Alfa-2b + Ribavirin
Number analyzed (Participants) | 2312 | 496 | 292 | 93 | 821 | 86
percentage of participants | 60.3 | 65.7 | 76.7 | 88.2 | 90.7 | 87.2

ADVERSE EVENTS:
Time Frame: Up to 118 weeks
Description: An AE was defined as any adverse medical event that occurred after the participant used the investigational medicinal product (IMP) or other intervention behaviors specified by the protocol in the clinical trial regardless of relationship to the study treatment.
Arm/Group | Dual Therapy: Peg-IFN Alfa-2a + Ribavirin | Dual Therapy: Peg-IFN Alfa-2b + Ribavirin | Triple Therapy: Boceprevir + Peg-IFN Alfa-2a + Ribavirin | Triple Therapy: Boceprevir + Peg-IFN Alfa-2b + Ribavirin | Triple Therapy: Telaprevir + Peg-IFN Alfa-2a + Ribavirin | Triple Therapy: Telaprevir + Peg-IFN Alfa-2b + Ribavirin
Serious Adverse Events (participants affected / at risk) | 148/2312 | 33/496 | 43/292 | 9/93 | 163/821 | 4/86
Other Adverse Events (participants affected / at risk) | 1225/2312 | 287/496 | 207/292 | 79/93 | 709/821 | 72/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dual Therapy: Peg-IFN Alfa-2a + Ribavirin (N=2312) | Dual Therapy: Peg-IFN Alfa-2b + Ribavirin (N=496) | Triple Therapy: Boceprevir + Peg-IFN Alfa-2a + Ribavirin (N=292) | Triple Therapy: Boceprevir + Peg-IFN Alfa-2b + Ribavirin (N=93) | Triple Therapy: Telaprevir + Peg-IFN Alfa-2a + Ribavirin (N=821) | Triple Therapy: Telaprevir + Peg-IFN Alfa-2b + Ribavirin (N=86)
Acquired haemophilia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Agranulocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 25 | 2 | 9 | 3 | 57 | 1
Aplasia pure red cell (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Haemolysis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 2 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 12 | 1 | 4 | 0 | 2 | 0
Pancytopenia (Blood and lymphatic system disorders) | 5 | 0 | 0 | 1 | 5 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 2 | 2 | 1 | 4 | 0
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Angina unstable (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Atrioventricular block (Cardiac disorders) | 1 | 0 | 1 | 0 | 0 | 0
Bundle branch block left (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 1 | 0 | 4 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cardiovascular insufficiency (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1 | 1 | 0 | 1 | 0
Coronary artery occlusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 1 | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Tricuspid valve incompetence (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cerebrovascular arteriovenous malformation (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1 | 0
Deafness (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 1 | 1 | 0 | 0 | 0 | 0
Thyroiditis (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0
Blindness unilateral (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Eye oedema (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Retinal detachment (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Retinal vein thrombosis (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Retinopathy (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Visual acuity reduced (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 2 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Alcoholic pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 2 | 1 | 1 | 0 | 1 | 0
Chronic gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Gastric ulcer perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 2 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Reflux gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Varices oesophageal (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 3 | 1
Asthenia (General disorders) | 1 | 0 | 0 | 0 | 1 | 1
Chest discomfort (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Death (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 2 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 6 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Oedema (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 2 | 0
Pyrexia (General disorders) | 1 | 1 | 1 | 1 | 3 | 0
Systemic inflammatory response syndrome (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Vascular stent restenosis (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 2 | 0 | 0 | 0 | 2 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 6 | 0
Hepatic failure (Hepatobiliary disorders) | 2 | 1 | 0 | 0 | 2 | 0
Hepatitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hepatocellular injury (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hepatorenal syndrome (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Abdominal abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Acinetobacter infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 3 | 0 | 0 | 0 | 0 | 0
Arthritis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Atypical mycobacterial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Brain abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Dermo-hypodermitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
End stage AIDS (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Endocarditis (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0
Enteritis infectious (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Erysipelas (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0
Escherichia sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Extradural abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0 | 3 | 0
Hepatitis B (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Infected dermal cyst (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Infectious pleural effusion (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Listeria sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0
Lung abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Meningitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Neutropenic sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0
Orchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Peritonitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Peritonitis bacterial (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0
Peritonsillar abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 12 | 2 | 1 | 0 | 6 | 0
Pulmonary sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 1 | 0 | 5 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 2 | 1 | 0 | 4 | 0
Septic arthritis staphylococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Septic shock (Infections and infestations) | 1 | 0 | 1 | 0 | 4 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Staphylococcal abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0
Streptococcal endocarditis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0
Tracheobronchitis mycoplasmal (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Tuberculosis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 5 | 1 | 0 | 0 | 2 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Cystitis radiation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Fractured sacrum (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 2 | 0
Pneumocephalus (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Skull fractured base (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Synovial rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
VIIIth nerve injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Alpha 1 foetoprotein increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Blood pressure increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Blood urea increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Cachexia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Tetany (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Neck mass (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Osteitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
B-cell lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Cardiac myxoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Hepatic cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 0 | 1 | 0 | 5 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Non-hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Papillary cystadenoma lymphomatosum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Complex partial seizures (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Diabetic encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Diabetic hyperglycaemic coma (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Facial paresis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hemiplegia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 1 | 1 | 0 | 0 | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Metabolic encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Occipital neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Optic neuritis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Sensorimotor disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 2 | 0
Toxic leukoencephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0 | 0 | 2 | 0
Wernicke's encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Acute psychosis (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2 | 0
Alcoholism (Psychiatric disorders) | 1 | 0 | 0 | 0 | 2 | 0
Bipolar disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 5 | 2 | 0 | 0 | 1 | 0
Irritability (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Mental disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Panic attack (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Persecutory delusion (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Somatoform disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0 | 1 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 5 | 0
Calculus ureteric (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Lupus nephritis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 3 | 1
Urethral stenosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Menometrorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 2 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 2 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0
Excessive granulation tissue (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 0 | 6 | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vascular purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Victim of homicide (Social circumstances) | 1 | 0 | 0 | 0 | 0 | 0
Polypectomy (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0 | 0
Aortic aneurysm (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 0 | 0 | 0 | 0 | 0
Hypertensive crisis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Peripheral venous disease (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Shock haemorrhagic (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Temporal arteritis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Venous thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Venous thrombosis limb (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dual Therapy: Peg-IFN Alfa-2a + Ribavirin (N=2312) | Dual Therapy: Peg-IFN Alfa-2b + Ribavirin (N=496) | Triple Therapy: Boceprevir + Peg-IFN Alfa-2a + Ribavirin (N=292) | Triple Therapy: Boceprevir + Peg-IFN Alfa-2b + Ribavirin (N=93) | Triple Therapy: Telaprevir + Peg-IFN Alfa-2a + Ribavirin (N=821) | Triple Therapy: Telaprevir + Peg-IFN Alfa-2b + Ribavirin (N=86)
Anaemia (Blood and lymphatic system disorders) | 435 | 141 | 112 | 42 | 351 | 43
Neutropenia (Blood and lymphatic system disorders) | 258 | 64 | 35 | 25 | 84 | 24
Leukopenia (Blood and lymphatic system disorders) | 129 | 47 | 8 | 6 | 59 | 31
Thrombocytopenia (Blood and lymphatic system disorders) | 138 | 26 | 31 | 5 | 94 | 23
Asthenia (General disorders) | 236 | 72 | 53 | 23 | 245 | 8
Fatigue (General disorders) | 244 | 53 | 68 | 23 | 170 | 13
Influenza like illness (General disorders) | 167 | 38 | 31 | 17 | 97 | 7
Pyrexia (General disorders) | 147 | 45 | 13 | 10 | 33 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 160 | 55 | 37 | 16 | 240 | 10
Rash (Skin and subcutaneous tissue disorders) | 85 | 25 | 24 | 9 | 155 | 9
Insomnia (Psychiatric disorders) | 121 | 40 | 18 | 7 | 100 | 4
Depression (Psychiatric disorders) | 82 | 32 | 15 | 8 | 70 | 3
Decreased appetite (Metabolism and nutrition disorders) | 101 | 47 | 25 | 16 | 118 | 8
Headache (Nervous system disorders) | 102 | 39 | 33 | 15 | 94 | 5
Weight decreased (Investigations) | 97 | 28 | 14 | 9 | 47 | 1
Nausea (Gastrointestinal disorders) | 85 | 30 | 36 | 24 | 134 | 11
Dry skin (Skin and subcutaneous tissue disorders) | 51 | 11 | 22 | 10 | 66 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 69 | 20 | 14 | 10 | 51 | 2
Diarrhoea (Gastrointestinal disorders) | 59 | 8 | 17 | 11 | 78 | 4
Anal pruritus (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 61 | 4
Vomiting (Gastrointestinal disorders) | 26 | 9 | 8 | 5 | 47 | 6
Haemorrhoids (Gastrointestinal disorders) | 9 | 1 | 5 | 2 | 47 | 6
Abdominal pain (Gastrointestinal disorders) | 32 | 2 | 10 | 6 | 39 | 0
Dry mouth (Gastrointestinal disorders) | 21 | 3 | 7 | 4 | 27 | 5
Irritability (Psychiatric disorders) | 48 | 7 | 10 | 4 | 49 | 1
Dysgeusia (Nervous system disorders) | 13 | 5 | 33 | 14 | 40 | 1
Dizziness (Nervous system disorders) | 40 | 19 | 9 | 8 | 24 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 103 | 23 | 23 | 10 | 72 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 54 | 16 | 18 | 9 | 72 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 10 | 4 | 5 | 5 | 9 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 45 | 19 | 18 | 6 | 53 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 76 | 19 | 8 | 8 | 53 | 3
Haemoglobin decreased (Investigations) | 22 | 9 | 1 | 0 | 16 | 13
Neutrophil count increased (Investigations) | 6 | 1 | 0 | 0 | 7 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.